CLINICAL TRIAL: NCT00607620
Title: Disseminating Organizational SBI Services (DO-SBIS) at Trauma Centers
Brief Title: Disseminating Organizational SBI Services at Trauma Centers
Acronym: DO-SBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Harborview Injury Prevention and Research Center (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30660; 1R01AA016102-01 (NIH)
Record Dates: First submitted 2008-01-29; First posted 2008-02-06 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Alcohol Abuse; Alcohol Dependence
Keywords: Alcohol Abuse; Alcohol Dependence; Alcohol Use Disorder; Screening; Brief Intervention; Motivational Interviewing
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Providers receive training in alcohol screening and brief interventions from study staff in compliance with American College of Surgeons' Alcohol Screening and Brief Intervention Mandate
  Interventions: Behavioral: Brief Intervention
- Usual Care (No Intervention): Usual care for alcohol use problems after American College of Surgeons' Alcohol Screening and Brief Intervention Mandate

INTERVENTIONS:
Behavioral: Brief Intervention — Training in brief interventions for alcohol use disorders, with a focus on motivational interviewing
  Other Names: Motivational Interviewing
  Arms: Intervention

SUMMARY:
The goal of the Disseminating Organizational Screening and Brief Interventions Services (DO-SBIS) investigation is to capitalize on the unique opportunity afforded by the American College of Surgeons' mandate by taking early steps to insure high quality, evidence-based SBI services are implemented and outcomes are assessed. In the first phase of the investigation, SBI services will be assessed for all 190 level I trauma centers in the United States. In the second phase of the investigation, 20 level I trauma centers will be selected for randomization to intervention or control conditions.

DETAILED DESCRIPTION:
Each year in the United States approximately 2.5 million individuals are so severely injured that they require inpatient hospital admission. The integration of screening and brief interventions (SBI) into acute injury care has the potential to markedly increase the number of patients who receive needed services and has been a longstanding public health objective. In January of 2005 the American College of Surgeons, the primary agency responsible for developing trauma center requirements, passed a landmark resolution mandating that level I trauma centers must screen injured patients for an alcohol use disorder, and provide an intervention to those who screen positive. Preliminary studies suggest that there is a substantial risk that the SBI mandate will be implemented with marked variability and that low quality SBI procedures could become the default standard of trauma center care.

Providers at each intervention trauma center will receive workshop training and ongoing telephone coaching in the delivery of evidence-based motivational interviewing (MI) intervention; MI training will be embedded within evidence-based organizational development activities that aim to facilitate the integration of SBI services into routine trauma center care. Control trauma centers will implement SBI care as usual. The investigation hypothesizes that intervention trauma centers, when compared to control trauma centers, will demonstrate higher quality SBI, as evidenced by greater provider proficiency in SBI delivery, significant reductions in 6- and 12-month post-injury alcohol use in patients receiving SBI, and enhanced organizational acceptance of SBI services. Without DO-SBIS baseline data on SBI services and follow-up RCT data on patient, provider, and organizational outcomes, a critical opportunity to provide empiric support of a historic policy decision to require alcohol services at level I trauma centers could be lost. The DO-SBIS interdisciplinary research group includes trauma surgery opinion leaders who are dedicated to implementing future policy mandates that derive from the DO-SBIS research program. Future mandates will aim to strengthen and refine trauma center delivery of evidence-based SBI services. The dissemination of high quality SBI services at level I trauma centers has the potential to influence alcohol policy in other health care settings nationwide.

ELIGIBILITY:
Inclusion Criteria:

* For provider subjects: staff at trauma centers selected by study
* For patient subjects: admitted to trauma centers selected by study, positive blood alcohol levels, able to provide two follow-up contacts

Exclusion Criteria:

* For Providers: Once a trauma center is selected for participation, providers will be selected from existing hospital staff.
* For Patients: Patients so severely injured that they cannot participate in study procedures will be excluded;
* Patients who are admitted after self-inflicted injury, or are psychotic and therefore require more intensive acute interventions, will not be included in the study;
* Injured hospitalized prisoners are excluded.
* Children under the age of 18 are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas F Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Zatzick D, Donovan DM, Jurkovich G, Gentilello L, Dunn C, Russo J, Wang J, Zatzick CD, Love J, McFadden C, Rivara FP. Disseminating alcohol screening and brief intervention at trauma centers: a policy-relevant cluster randomized effectiveness trial. Addiction. 2014 May;109(5):754-65. doi: 10.1111/add.12492. Epub 2014 Feb 28. PMID 24450612
- [Derived] Zatzick D, Palinkas L, Chambers DA, Whiteside L, Moloney K, Engstrom A, Prater L, Russo J, Wang J, Abu K, Iles-Shih M, Bulger E. Integrating pragmatic and implementation science randomized clinical trial approaches: a PRagmatic Explanatory Continuum Indicator Summary-2 (PRECIS-2) analysis. Trials. 2023 Apr 21;24(1):288. doi: 10.1186/s13063-023-07313-0. PMID 37085877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 409 | 469
Completed | 409 | 469
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 409 | 469 | 878
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (14.7) | 36.4 (14.0) | 36.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 103 | 208
  Male | 304 | 366 | 670
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Baseline: White | 253 | 292 | 545
  Baseline: Black or African American | 62 | 63 | 125
  Baseline: American Indian or Alaska Native | 25 | 13 | 38
  Baseline: Asian | 8 | 6 | 14
  Baseline: Hispanic | 61 | 95 | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hazardous Drinking
Description: The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) as a dichotomous measure. AUDIT Scores of ≥8 for men and ≥5 for women indicate hazardous drinking.
Time Frame: The investigators will assess at baseline, 6-month and 12-month.
Population: Overall number of participants analyzed differs from the number of participants analyzed in Month 6 and Month 12 due to lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 409 | 469
Participants
  Baseline | 292 | 309
  Month 6: number analyzed (Participants) | 326 | 378
  Month 6 | 201 | 223
  Month 12: number analyzed (Participants) | 292 | 332
  Month 12 | 166 | 198
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.79 to 0.98]

2. Primary Outcome: Alcohol Use Problems
Description: The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) as a continuous measure. The 10-item scale score ranges from 0-40, with higher values indicating a worse outcome.
Time Frame: The investigators will assess at baseline, 6-month and 12-month.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 409 | 469
units on a scale
  Baseline | 10.5 (5.1) | 9.7 (4.9)
  Month 6: number analyzed (Participants) | 326 | 378
  Month 6 | 8.8 (6.3) | 8.5 (6.5)
  Month 12: number analyzed (Participants) | 292 | 332
  Month 12 | 8.2 (6.1) | 8.5 (6.3)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.1 to -0.3] — The data represented refers to the group mean difference (intervention versus control) of the change score between baseline to 12-months

3. Secondary Outcome: Number of Abstinent Days
Description: The investigators will use the Form 90 to assess the number of days within the last 90 days in which a patient did not consume alcohol.
Time Frame: The investigators will assess at 6- and 12-month.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 409 | 469
days
  Month 6: number analyzed (Participants) | 326 | 378
  Month 6 | 74.2 (1.35) | 73.4 (1.25)
  Month 12: number analyzed (Participants) | 292 | 332
  Month 12 | 75.5 (1.37) | 71.3 (1.27)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Net) = 3.4, 95% CI 2-sided [0.4 to 6.4] — The data represented refers to the group mean difference (intervention versus control) of the change score between 6-months and 12-months

4. Secondary Outcome: Number of Binge Drinking Days
Description: The investigators will use the Form 90 to assess the number of days in which a male participants consumed ≥5 alcoholic drinks and female participants consumed ≥4 alcoholic drinks
Time Frame: The investigators will assess at 6-month and 12-month.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 409 | 469
days
  Month 6: number analyzed (Participants) | 326 | 378
  Month 6 | 9.4 (1.14) | 10.6 (1.13)
  Month 12: number analyzed (Participants) | 292 | 332
  Month 12 | 9.4 (1.16) | 11.4 (1.10)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Net) = -0.7, 95% CI 2-sided [-3.3 to 1.9] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Alcohol Use Problems
Description: The investigators will use the Short Inventory of Problems (SIP) as a continuous measure. The 16-item scale score ranges from 0-48 with higher scores indicating worse outcomes.
Time Frame: The investigators will assess at 6-month and 12-month.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 409 | 469
units on a scale
  Month 6: number analyzed (Participants) | 326 | 378
  Month 6 | 3.3 (0.42) | 3.38 (0.39)
  Month 12: number analyzed (Participants) | 292 | 332
  Month 12 | 2.99 (0.43) | 3.08 (0.41)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Net) = -0.01, 95% CI 2-sided [-1.02 to 0.99] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 10/409 | 3/469
Serious Adverse Events (participants affected / at risk) | 1/409 | 1/469
Other Adverse Events (participants affected / at risk) | 62/409 | 65/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=409) | Usual Care (N=469)
Suicide Attempt (Psychiatric disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=409) | Usual Care (N=469)
Patient Health Questionnaire (PHQ-9) Score of >0 (Psychiatric disorders) | 62 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No